CLINICAL TRIAL: NCT02346149
Title: Effect of Acute Hyperglycemia on Renal Tissue Oxygenation as Measured By BOLD-MRI in Individuals With Impaired Glucose Tolerance and Controls
Brief Title: Effect of Acute Hyperglycemia on Renal Tissue Oxygenation
Acronym: Glucox
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Michel Burnier, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNSF132913
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hyperglycemia; Glucose Intolerance
MeSH Terms: conditions — Hyperglycemia; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: IV administration of 0.15 g/kg of glucose in a 20% solution under standard hydration and fasting conditions
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient with impaired glucose tolerance (Other): Bold-MRI before and after glucose injection
  Interventions: Other: glucose 20%

INTERVENTIONS:
Other: glucose 20% — Intravenous infusion (0.75 ml / kg) over 1 min

SUMMARY:
Diabetes Mellitus (DM) includes several metabolic diseases all characterized by high sugar levels in the blood. Although diabetic nephropathy is widespread, its underlying pathophysiological mechanisms remain poorly understood and, so far, little progress has been made to prevent the development of diabetic nephropathy and to delay kidney functions decline.

Increasing amount of data based on animal studies support the pathogenic role of tissue hypoxia in the development and progression of diabetic nephropathy. Blood Oxygenation-Level Dependent Magnetic Resonance Imaging (BOLD-MRI) is increasingly used in research to measure cortical and medullary oxygenation in a non-invasive manner. Interestingly, in two cross-sectional clinical studies, we have recently found a positive correlation between high circulating blood glucose levels and cortical R2* levels in type 2 DM patients. This discovery suggests that an increase in glycemia might acutely decrease renal tissue oxygenation.

The goal of this study is to investigate the impact of serum glucose on renal tissue oxygenation in healthy subjects and subjects with glucose intolerance.

DETAILED DESCRIPTION:
Therefore, we plan to recruit 10 healthy subjects and 10 glucose intolerant patients with preserved kidney functions and to perform repetitive BOLD-MRI, before and after the administration of IV glucose. This will allow us to study the influence of hyperglycemia as a single factor, regardless of inflammation, oxidative stress and medical treatments, such as oral hypoglycemic agents and/or insulin, which are confounding factors present in all DM patients.

The main hypothesis of the project is that acute hyperglycemia could be partially responsible for renal tissue hypoxia detected in diabetic nephropathy cases.

In this study we will include 60 participants with a family history of diabetes, with a Body Mass Index (BMI) over 25 kg / m2 and/or having glucose intolerance. Each participant will undergo an initial glucose tolerance test. In total, we will select 10 participants with impaired glucose tolerance and 10 healthy subjects (matched for sex and age), to be included as control group.

Selected subjects will return for a third visit at CHUV (V3): they will start at home with an oral hydration protocol (load dose of 3 ml / kg at 8:00 am, followed by 1 ml / kg every hour between 9:00 am and 3:00 pm to avoid as much as possible changes in kidney perfusion). Patients will arrive at the Department of Nephrology and Hypertension (CHUV) at 11.00 am. In this occasion, two catheters will be placed into each patient's arm. Later, participants will be escorted to the Radiology Department to undergo four renal oxygenation imaging (between 1:00 pm and 2:00 pm) by the mean of BOLD-MRI technique. During this period, patients and control subjects will lie down and are not allowed to stand up. At T0, they will receive a bolus (0.75 ml / kg) of glucose 20%. Subsequently, four BOLD-MRI scans, together with blood tests, will be performed at T0, T1 (+10 min), T2 (+20 min), T3 (+30 min). Sodium intake will be measured by 24 hours urinary collection the day before V3 (sodium is known to influence R2*).

ELIGIBILITY:
Inclusion Criteria:

* Positive family history of diabetes
* BMI > 25 kg / m2
* eGFR > 60 ml / min / 1.73 m2
* Understanding and signing the informed consent

Exclusion Criteria:

* Documented cardiac disease
* Documented liver failure
* Renal malformations, kidney diseases or documented renal artery stenosis
* History of organ transplantation
* Significant comorbidities compromising life expectancy
* Anemia
* Type 1 or 2 diabetes
* Psychiatric illness
* Contraindication to MRI
* Pregnancy or breastfeeding
* Chronic drug intake such as antihypertensive (except for beta blockers and calcium antagonists), non steroidal anti-inflammatory drugs, diuretics or oral antidiabetics
* Blood donation 2 months before the MRI investigation day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Cortical and medullary renal R2* MRI signal variation, before, during and after an induced hyperglycemic state | Four R2* imaging will be performed during an investigation day between 1:00 pm and 2:00 pm
Intergroup variability of MRI R2* signal, before, during and after an induced hyperglycemic state | Four R2* imaging will be performed during an investigation day between 1:00 pm and 2:00 pm

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Department of Nephrology, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Pruijm M, Hofmann L, Zanchi A, Maillard M, Forni V, Muller ME, Wuerzner G, Vogt B, Stuber M, Burnier M. Blockade of the renin-angiotensin system and renal tissue oxygenation as measured with BOLD-MRI in patients with type 2 diabetes. Diabetes Res Clin Pract. 2013 Feb;99(2):136-44. doi: 10.1016/j.diabres.2012.11.004. Epub 2012 Dec 14. PMID 23245807